CLINICAL TRIAL: NCT02399956
Title: Lactation Outcomes Among Survivors of Pediatric Cancer
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LACOUT
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Cancer; Leukemia
Keywords: Lactation; Pediatric malignancies; Cancer survivor
MeSH Terms: conditions — Neoplasms; Leukemia; Breast Feeding | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survivors: Participants will be recruited from the St. Jude Lifetime Cohort (SJLIFE protocol) and the After Completion of Therapy (ACT) Clinic at St. Jude Children's Research Hospital.
  Intervention: Survey
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Those who agree to participate will complete a cross-sectional survey on lactation outcomes (LACOUT). Eligible participants who consent to our study will complete the LACOUT questionnaire. The questionnaire uses the same breastfeeding measures as the CDC's Project First surveys and adds 21 items that are specific to the participant's cancer treatment and current health status.
  Other Names: Questionnaire

SUMMARY:
While the majority of women in the general population can breastfeed successfully, the investigators have limited knowledge about the correlates and sequelae of lactation success among women treated for pediatric malignancies. Childhood cancer treatments are known to cause late effects that frequently involve the endocrine system. Because normal lactation is dependent upon interplay of multiple endocrine factors, the investigators anticipate more breastfeeding difficulties in survivors that have diabetes, growth hormone deficiencies, thyroid disorders and obesity. In order to more fully inform clinicians and female survivors, the study of the burden of lactation failure is needed to begin to address the impact of pediatric cancer therapy on lactation success/failure and to examine the association of specific endocrine disorders on lactation outcomes.

DETAILED DESCRIPTION:
Participants will complete a cross-sectional survey. Responses will be compared with a national sample of healthy women from Project First (Infant Feeding Practices Survey II).

Primary Objective:

* To describe breastfeeding outcomes (intention, initiation, duration, and weaning) among female SJLIFE protocol participants 18 years of age and older who reported a live birth.

Secondary Objective:

* To compare breastfeeding outcomes between childhood cancer survivors and healthy mothers.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the SJLIFE protocol or patients in the After Completion of Therapy (ACT) Clinic, both at St. Jude Children's Research Hospital.
* Female
* 18 years of age or older
* At least one reported live birth after childhood cancer diagnosis and treatment.

Exclusion Criteria:

* Unable to read and write.
* Unable to read and understand English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females who are childhood cancer survivors and have reported at least one live birth after cancer diagnosis and treatment.
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of survivors who experience successful breastfeeding outcome by age at diagnosis | Once, at enrollment (Day 1)
Number of survivors who experience successful breastfeeding outcome by years since diagnosis | Once, at enrollment (Day 1)
  Years since diagnosis will equal the years since diagnosis prior to first pregnancy resulting in a live birth.
Number of survivors who experience successful breastfeeding outcome by therapy with radiation | Once, at enrollment (Day 1)
Number of survivors who experience successful breastfeeding outcome by therapy with surgery | Once, at enrollment (Day 1)
  Includes chest and/or brain surgery.
Number of survivors who experience successful breastfeeding outcome by diagnosis of growth hormone deficiency | Once, at enrollment (Day 1)
  Growth hormone deficiency indicated by low IGF-1
Number of survivors who experience successful breastfeeding outcome by diagnosis of hypothyroidism | Once, at enrollment (Day 1)
  Hypothyroidism, primary or central, measured by TSH level.
Number of survivors who experience successful breastfeeding outcome by diagnosis of diabetes mellitus | Once, at enrollment (Day 1)
Number of survivors who experience successful breastfeeding outcome by diagnosis of obesity | Once, at enrollment (Day 1)
  Obesity (BMI) prior to pregnancy.

SECONDARY OUTCOMES:
Number of survivors who experience successful breastfeeding outcome compared to healthy women | Once, at enrollment (Day 1)
  Breastfeeding outcomes (intention, initiation, and duration/weaning) will be determined by self-report, and dichotomized for analysis. Intention is defined as a mother's specific plan to breastfeed her infant prior to birth (yes/no); initiation is defined as ever having started breastfeeding (yes/no); duration is defined as at least 6 months of breastfeeding (yes/no); and weaning is defined as breastfeeding cessation after 1 year (yes/no).
  Data from survivors will be compared with a national sample of healthy women (n=2,000) who responded to the Project First survey (2009). The Infant Feeding Practices Survey II (Project First) is a longitudinal study developed by the Food and Drug Administration and the Centers for Disease Control and Prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Cox, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Ogg S, Klosky JL, Chemaitilly W, Srivastava DK, Wang M, Carney G, Ojha R, Robison LL, Cox CL, Hudson MM. Breastfeeding practices among childhood cancer survivors. J Cancer Surviv. 2020 Aug;14(4):586-599. doi: 10.1007/s11764-020-00882-y. Epub 2020 Apr 14. PMID 32291564
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols